CLINICAL TRIAL: NCT05399628
Title: LISA Catheter With Marked vs. Unmarked Tip in Extremely Low Birth Weight Infants With RDS: a Crossover Randomized Controlled Manikin Trial
Brief Title: LISA Catheter With Marked vs. Unmarked Tip in Extremely Low Birth Weight Infants With RDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEOUNIPD2(2022)
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Intervention Model Description: Participants in AB arm will be assigned to perform the procedure with LISA catheter with marked tip, followed by the procedure with LISA catheter with unmarked tip. Participants in BA arm will be assigned to the reverse sequence. A washout period of 6 hours (one procedure in the morning and one in the afternoon) will be included to reduce any carryover effect
Masking Description: Due to the characteristics of the intervention, both participants and outcome assessors cannot be masked. The statistician will be blind to the intervention arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surfactant administration with less invasive surfactant administration (LISA) marked tip catheter (Experimental): Participants will be assigned to perform the procedure with a LISA catheter with a marked tip
  Interventions: Device: Surfactant administration with less invasive surfactant administration (LISA) marked tip catheter
- Surfactant administration with less invasive surfactant administration (LISA) unmarked tip catheter (Active Comparator): Participants will be assigned to perform the procedure with a LISA catheter with an unmarked tip
  Interventions: Device: Surfactant administration with less invasive surfactant administration (LISA) unmarked tip catheter

INTERVENTIONS:
Device: Surfactant administration with less invasive surfactant administration (LISA) marked tip catheter — Participants will be assigned to perform the procedure with LISA catheter with a marked tip
  Arms: Surfactant administration with less invasive surfactant administration (LISA) marked tip catheter
Device: Surfactant administration with less invasive surfactant administration (LISA) unmarked tip catheter — Participants will be assigned to perform the procedure with LISA catheter with an unmarked tip
  Arms: Surfactant administration with less invasive surfactant administration (LISA) unmarked tip catheter

SUMMARY:
This is an unblinded, randomized, controlled, crossover (AB/BA) trial of surfactant treatment with LISA catheter with a marked tip vs. LISA catheter with an unmarked tip in a manikin simulating an extremely low birth weight infant. Participants will be level III NICU consultants and residents. Randomization will be performed using a computer-generated random assignment list. The primary outcome measure will be the positioning of the device at the correct depth in the trachea. The secondary outcome measures will be the time and number of attempts to achieve the correct depth and participant satisfaction.

DETAILED DESCRIPTION:
Although less invasive surfactant administration (LISA) offers some advantages in ventilation procedure and neonatal outcomes, achieving the correct depth in the trachea using a LISA catheter may be difficult. This may have some drawbacks such as impaired surfactant administration (reducing the efficacy of the procedure) or prolonged duration of the laryngoscopy (aggravating the invasiveness of the procedure).

The aims of the present study should be: i) positioning of the device at the correct depth in the trachea, ii) time and number of attempts to achieve the correct depth, iii) participant satisfaction.

This is an unblinded, randomized, controlled, crossover (AB/BA) trial of surfactant treatment with LISA catheter with a marked tip vs. LISA catheter with an unmarked tip in a manikin simulating an extremely low birth weight infant. Participants will be level III NICU consultants and residents. Randomization will be performed using a computer-generated random assignment list. The primary outcome measure will be the positioning of the device at the correct depth in the trachea. The secondary outcome measures will be the time and number of attempts to achieve the correct depth and participant satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Level III NICU consultants and residents will be eligible to participate in the study

Exclusion Criteria:

* Refusal to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Number of participants who will achieve the positioning of the device at the correct depth in the trachea | 5 minutes
  Number of participants who will achieve the positioning of the device at the correct depth in the trachea (as assessed by the external observer using a laryngoscope).

SECONDARY OUTCOMES:
Time for positioning the device in the trachea | 5 minutes
  The time of device positioning will be defined as the time elapsed from the positioning of the laryngoscope in the manikin mouth to the connection of the syringe to the catheter
Number of attempts for positioning the device in the trachea | 5 minutes
  The total number of attempts for positioning the device in the trachea
Participant opinion on using the device | 10 minutes
  Participant opinion on using the device which will be evaluated using a Likert scale (1 worse outcome to 5 best outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Daniele Trevisanuto, Padua, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon motivated request to the corresponding author
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433